CLINICAL TRIAL: NCT06792370
Title: Effectiveness of an Alternative Protocol in the Management of Acute Malnutrition in Children Aged 6-59 Months in Burkina Faso: Reduced Dose of RUTF for SAM Children and RUTF Instead of RUSF for MAM Children
Brief Title: Effectiveness of an Alternative Protocol in the Management of Acute Malnutrition
Acronym: Alternat-MAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INV-016380-2
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Malnutrition with No Complications
Keywords: Effectiveness; acute malnutrition; management; treatment; reduced dose; Ready-to-Use Supplementary Foods; Ready-to-Use Therapeutic Foods; uncomplicated; without complication
MeSH Terms: interventions — Sarcoglycans

STUDY DESIGN:
Intervention Model Description: Individually randomized and controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- MAM RUTF (Experimental): Participants with MAM in this arm will receive a dose of 500 kcal/kg/day of RUTF
  Interventions: Dietary Supplement: ready-to-use therapeutic food (for children with MAM)
- MAM RUSF (Active Comparator): Participants with MAM in this arm will receive a dose of 540 kcal/kg/day of RUSF
  Interventions: Dietary Supplement: Ready-to-use supplementary food
- SAM Reduced-dose RUTF 1 (R-RUTF 1) (Experimental): Participants with SAM in this arm will receive a dose of 150-185 kcal/kg/day of RUTF until programmatic recovery
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food - Reduced dose 1
- SAM Reduced-dose RUTF 2 (R-RUTF 2) (Experimental): Participants with SAM in this arm will receive a dose of 150-185 kcal/kg/day of RUTF until the child is no longer severely malnourished and does not have nutritional oedema then 100-130 kcal/kg/day of RUTF until programmatic recovery
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food - Reduced dose 2
- SAM standard dose RUTF (S-RUTF) (Active Comparator): Participants with SAM in this arm will receive the standard dose of RUTF according to the national protocol for the integrated management of acute malnutrition in Burkina Faso
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food - Standard dose

INTERVENTIONS:
Dietary Supplement: ready-to-use therapeutic food (for children with MAM) — Each child with MAM will be supplemented with RUTF for a maximum of 12 weeks. He/she will be followed subsequently up to 24 weeks.
  Other Names: RUTF
  Arms: MAM RUTF
Dietary Supplement: Ready-to-use supplementary food — Each child with MAM will be supplemented with RUSF for a maximum of 12 weeks. He/she will be followed subsequently up to 24 weeks post recovery
  Other Names: RUSF
  Arms: MAM RUSF
Dietary Supplement: Ready to Use Therapeutic Food - Reduced dose 1 — Each child with SAM will be treated with a reduced dose for a maximum of 12 weeks : dose of 150-185 kcal/kg/day of RUTF until programmatic recovery. He/she will be followed subsequently up to 24 weeks post recovery.
  Other Names: R-RUTF 1
  Arms: SAM Reduced-dose RUTF 1 (R-RUTF 1)
Dietary Supplement: Ready to Use Therapeutic Food - Standard dose — Each child with SAM will be treated with a standard dose (according to the national protocol for the integrated management of acute malnutrition in Burkina Faso) for a maximum of 12 weeks. He/she will be followed subsequently up to 24 weeks post recovery.
  Other Names: S-RUTF
  Arms: SAM standard dose RUTF (S-RUTF)
Dietary Supplement: Ready to Use Therapeutic Food - Reduced dose 2 — Each child with SAM will be treated with a reduced dose for a maximum of 12 weeks : dose of 150-185 kcal/kg/day of RUTF until the child is no longer severely malnourished and does not have nutritional oedema then 100-130 kcal/kg/day of RUTF until programmatic recovery. He/she will be followed subsequently up to 24 weeks post recovery.
  Other Names: R-RUTF 2
  Arms: SAM Reduced-dose RUTF 2 (R-RUTF 2)

SUMMARY:
This experimental study aims to test an alternative protocol for managing acute malnutrition in children aged 6-59 months in Burkina Faso. This alternative protocol consists of using RUTF instead of RUSF for the management of moderate acute malnutrition and reduced-dose RUTF instead of standard-dose RUTF for the treatment of severe acute malnutrition.

The main questions are:

1. Does treating children with moderate acute malnutrition using RUTF lead to a non-inferior programmatic and sustained recovery rate compared to the standard care with RUSF?
2. Does treating children with uncomplicated severe acute malnutrition using a reduced dose of RUTF lead to a non-inferior programmatic and sustained recovery rate compared to the standard care with a standard dose of RUFT?

Secondly, the study will investigate the effect of this alternative protocol compared to the standard protocol on cost-effectiveness, psychomotor development, weight and linear growth and incidence of relapses.

DETAILED DESCRIPTION:
In this trial, children presenting at the health center and fulfilling the inclusion criteria will be randomly allocated into one of the study groups in a ratio of 1:1:1 for severe acute malnutrition (SAM) without complication and 1:1 for moderate acute malnutrition (MAM).

Supplementation will be daily according to the child's weight for a maximum of 12 weeks, at which point the programmatic recovery assessment will be done. Those who recovered before or at this point will be subsequently followed up monthly for up to 3 months for sustained recovery assessment.

Follow-up visits will be done at the health center every week for children with SAM and every two weeks for children with MAM.

At each visit, anthropometric measurements will be performed; a morbidity questionnaire will be administered before the mother/caregiver receives the ration for the following period. For the measurement of adherence, mothers will be asked to bring back empty and unused sachets/packaging of supplements from the last visit. Questions will also be asked to the mother/caregiver on the difficulties encountered during consumption and the adverse events observed following the consumption of the supplements.

The evaluation of the psychomotor development will be performed in a subsample.

ELIGIBILITY:
1. MAM

   Inclusion Criteria:
   * Anthropometric measures:

     * (115 mm ≤ MUAC< 125 mm and -3 SDs ≤ WLZ < -2 SDs) OR
     * (115 mm ≤ MUAC< 125 mm and WLZ ≥ -2 SDs) OR
     * (MUAC ≥ 125 mm and -3 SDs ≤ WLZ < -2 SDs).
   * Age: 6 to 59 months
   * Parents' acceptance of biweekly visits until programme discharge and monthly visits for the post-programme follow up

   Exclusion Criteria:
   * Failure of appetite test
   * Medical complications requiring hospital treatment
   * Presence of any congenital anomaly or underlying chronic disease that may affect growth or the risk of infection
   * Presence of bilateral oedema
   * History of allergies to peanuts, milk, or soya
   * Relapse from MAM treatment or transfer from SAM treatment
   * Children who have recently (<2 months) taken part in a nutrition programme;
   * Residence outside the study area
   * Mother or caregivers deemed unable to comply with the necessary requirements of the study (particular medical condition of the mother or caregivers, etc.)
2. SAM

Inclusion Criteria:

* Anthropometric measures MUAC< 115 mm or WLZ< - 3 SDs;
* Age: 6-59 months;
* Parents' acceptance of weekly visits until programme discharge and monthly visits for the post-programme follow up.

Exclusion Criteria:

* Failure of appetite test
* Medical complications requiring hospital treatment
* Presence of any congenital anomaly or underlying chronic disease that may affect growth or the risk of infection
* Presence of bilateral oedema
* History of allergies to peanuts, milk or soya
* Relapse from MAM treatment or transfer from SAM treatment
* Children who have recently (<2 months) taken part in a nutrition programme;
* Residence outside the study area;
* Mother or caregivers deemed unable to comply with the necessary requirements of the study (particular medical condition of the mother or caregivers, etc.)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3521 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of programmatic recovery | From enrollment to the end of treatment (maximum 12 weeks)
  Number of children with a MUAC ≥ 125 mm and WLZ≥ -2 standard deviations for two consecutive visits at or before twelve (12) weeks since admission to the supplementation program in an arm divided by total number of children enrolled in the arm
Rate of sustained recovery | from programmatic recovery to 3 months after
  Number of children who maintain a MUAC ≥ 125 mm and WLZ≥ -2 SDs three (03) months after the programmatic recovery in an arm divided by total number of children with a programmatic recovery in the arm

SECONDARY OUTCOMES:
Cost per child treated | From enrollment to the end of treatment (maximum 12 weeks)
  Economic metric obtained by dividing the total costs for an arm by the number of children who received treatment in this arm
Cost per child recovered | From enrollment to the end of treatment (maximum 12 weeks)
  Economic metric obtained by dividing the total costs for an arm by the number of children recovered in this arm
Score of the extended version of Developmental Milestones Checklist (DMC-II) | Three points : enrollment , exit of the supplementation program (up to 12 weeks) and exit of the study (3 months after recovery)
  Psychomotor development of children aged 6-23 months will be assessed by a tool adapted for sub-Saharan Africa countries settings : the extended version of Developmental Milestones Checklist (DMC-II). DMC-II have 76 items and each item is scored from 0 to 2 :zero if the child has not yet started doing the skill, one if the child has been able to perform the skill in the past four weeks but not continually, two if the child has been able to perform the skill for the past four weeks continually. Thus, the minimum value of this score is 0 (indicating no developmental milestones achieved) and the maximum is 152 (full developmental milestones achieved).Higher scores indicate better developmental outcomes, reflecting more advanced motor, language, and personal-social skills.
Daily weight gain | From enrollment to the exit of the supplementation programme (maximum 12 weeks)]
  Refers to the increase in weight during the study period and is obtained by dividing the total weight gain in kilogram by the number of days since admission to the exit of the programme
Daily length gain | [Time Frame: From enrollment to the exit of the supplementation programme (maximum 12 weeks)
  Refers to the increase in length during the study period and is obtained by dividing the total length gain in centimetre by the number of days since admission to the exit of the supplementation programme (maximum 12 weeks)
Energy intake | From enrollment to the exit of the supplementation programme (maximum 12 weeks)
  Daily average of calories per kilogram obtained from the 24-hour recall
Rate of relapses | from programmatic recovery to 3 months after
  Number of children who return malnourished after programmatic recovery divided by the number of children with programmatic recovery
Length of stay | From enrollment to the exit of the supplementation programme (maximum 12 weeks)
  Duration in days from admission to programmatic recovery
Rate of defaulted | From enrollment to the exit of the supplementation programme (maximum 12 weeks)
  Number of children absent for three (3) consecutive visits in an arm divided of total number of children enrolled in the arm
Rate of treatment failure | From enrollment to the end of treatment (maximum 12 weeks)
  Number of participants with no weight gain after 5 weeks or at the third visit OR weight loss for more than 4 weeks in the program or at the second visit OR weight loss of more than 5% of body weight compared to admission weight at any time OR failure to meet discharge criteria after 3 months in an arm divided by total number of children enrolled in the arm
Number of adverse events | From enrollment to the exit of the supplementation programme (maximum 12 weeks)
  Number of incidents in which the use of the dietary supplement or data collection procedures is suspected to have contributed. This can be a physical event (e.g., a rash); a laboratory event (e.g., elevated blood sugar), or an increase in the severity or frequency of a pre-existing symptom or condition

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé, Ouagadougou, KADIOGO, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang CY, Trehan I, Wang RJ, Thakwalakwa C, Maleta K, Deitchler M, Manary MJ. Children successfully treated for moderate acute malnutrition remain at risk for malnutrition and death in the subsequent year after recovery. J Nutr. 2013 Feb;143(2):215-20. doi: 10.3945/jn.112.168047. Epub 2012 Dec 19. PMID 23256140
- [Background] Bailey J, Lelijveld N, Khara T, Dolan C, Stobaugh H, Sadler K, Lino Lako R, Briend A, Opondo C, Kerac M, Myatt M. Response to Malnutrition Treatment in Low Weight-for-Age Children: Secondary Analyses of Children 6-59 Months in the ComPAS Cluster Randomized Controlled Trial. Nutrients. 2021 Mar 24;13(4):1054. doi: 10.3390/nu13041054. PMID 33805040
- [Background] Maru Y, Tamiru D, Baye K, Chitekwe S, Laillou A, Darsene H, Abdulai R, Worku M, Belachew T. Effect of a simplified approach on recovery of children 6-59 months with wasting in Ethiopia: A noninferiority, cluster randomized controlled trial. Matern Child Nutr. 2024 Oct;20(4):e13670. doi: 10.1111/mcn.13670. Epub 2024 May 27. PMID 38800892
- [Background] Singh AS, Kang G, Ramachandran A, Sarkar R, Peter P, Bose A. Locally made ready to use therapeutic food for treatment of malnutrition a randomized controlled trial. Indian Pediatr. 2010 Aug;47(8):679-86. doi: 10.1007/s13312-010-0100-8. PMID 20972285
- [Background] Nackers F, Broillet F, Oumarou D, Djibo A, Gaboulaud V, Guerin PJ, Rusch B, Grais RF, Captier V. Effectiveness of ready-to-use therapeutic food compared to a corn/soy-blend-based pre-mix for the treatment of childhood moderate acute malnutrition in Niger. J Trop Pediatr. 2010 Dec;56(6):407-13. doi: 10.1093/tropej/fmq019. Epub 2010 Mar 23. PMID 20332221
- [Background] Medoua GN, Ntsama PM, Ndzana AC, Essa'a VJ, Tsafack JJ, Dimodi HT. Recovery rate of children with moderate acute malnutrition treated with ready-to-use supplementary food (RUSF) or improved corn-soya blend (CSB+): a randomized controlled trial. Public Health Nutr. 2016 Feb;19(2):363-70. doi: 10.1017/S1368980015001238. Epub 2015 May 5. PMID 25939394
- [Background] LaGrone LN, Trehan I, Meuli GJ, Wang RJ, Thakwalakwa C, Maleta K, Manary MJ. A novel fortified blended flour, corn-soy blend "plus-plus," is not inferior to lipid-based ready-to-use supplementary foods for the treatment of moderate acute malnutrition in Malawian children. Am J Clin Nutr. 2012 Jan;95(1):212-9. doi: 10.3945/ajcn.111.022525. Epub 2011 Dec 14. PMID 22170366
- [Background] Griswold SP, Langlois BK, Shen Y, Cliffer IR, Suri DJ, Walton S, Chui K, Rosenberg IH, Koroma AS, Wegner D, Hassan A, Manary MJ, Vosti SA, Webb P, Rogers BL. Effectiveness and cost-effectiveness of 4 supplementary foods for treating moderate acute malnutrition: results from a cluster-randomized intervention trial in Sierra Leone. Am J Clin Nutr. 2021 Sep 1;114(3):973-985. doi: 10.1093/ajcn/nqab140. PMID 34020452
- [Background] Karakochuk C, van den Briel T, Stephens D, Zlotkin S. Treatment of moderate acute malnutrition with ready-to-use supplementary food results in higher overall recovery rates compared with a corn-soya blend in children in southern Ethiopia: an operations research trial. Am J Clin Nutr. 2012 Oct;96(4):911-6. doi: 10.3945/ajcn.111.029744. Epub 2012 Sep 5. PMID 22952175
- [Background] Ackatia-Armah RS, McDonald CM, Doumbia S, Erhardt JG, Hamer DH, Brown KH. Malian children with moderate acute malnutrition who are treated with lipid-based dietary supplements have greater weight gains and recovery rates than those treated with locally produced cereal-legume products: a community-based, cluster-randomized trial. Am J Clin Nutr. 2015 Mar;101(3):632-45. doi: 10.3945/ajcn.113.069807. Epub 2015 Jan 7. PMID 25733649
- [Background] Javan R, Kooshki A, Afzalaghaee M, Aldaghi M, Yousefi M. Effectiveness of supplementary blended flour based on chickpea and cereals for the treatment of infants with moderate acute malnutrition in Iran: A randomized clinical trial. Electron Physician. 2017 Dec 25;9(12):6078-6086. doi: 10.19082/6078. eCollection 2017 Dec. PMID 29560163
- [Background] Nikiema L, Huybregts L, Kolsteren P, Lanou H, Tiendrebeogo S, Bouckaert K, Kouanda S, Sondo B, Roberfroid D. Treating moderate acute malnutrition in first-line health services: an effectiveness cluster-randomized trial in Burkina Faso. Am J Clin Nutr. 2014 Jul;100(1):241-9. doi: 10.3945/ajcn.113.072538. Epub 2014 May 7. PMID 24808482
- [Background] Daures M, Phelan K, Issoufou M, Kouanda S, Sawadogo O, Issaley K, Cazes C, Seri B, Ouaro B, Akpakpo B, Mendiboure V, Shepherd S, Becquet R. New approach to simplifying and optimising acute malnutrition treatment in children aged 6-59 months: the OptiMA single-arm proof-of-concept trial in Burkina Faso. Br J Nutr. 2020 Apr 14;123(7):756-767. doi: 10.1017/S0007114519003258. Epub 2019 Dec 10. PMID 31818335
- [Background] Stephenson KB, Agapova SE, Hendrixson DT, Koroma AS, Manary MJ. An Optimized Dose of Therapeutic Feeding Results in Noninferior Growth in Midupper Arm Circumference Compared with a Standard Dose in Children in Sierra Leone Recovering from Acute Malnutrition. Curr Dev Nutr. 2021 Feb 2;5(2):nzab007. doi: 10.1093/cdn/nzab007. eCollection 2021 Feb. PMID 33659773
- [Background] James PT, Van den Briel N, Rozet A, Israel AD, Fenn B, Navarro-Colorado C. Low-dose RUTF protocol and improved service delivery lead to good programme outcomes in the treatment of uncomplicated SAM: a programme report from Myanmar. Matern Child Nutr. 2015 Oct;11(4):859-69. doi: 10.1111/mcn.12192. Epub 2015 Apr 7. PMID 25850698
- [Background] Cazes C, Phelan K, Hubert V, Boubacar H, Bozama LI, Sakubu GT, Senge BB, Baya N, Alitanou R, Kouame A, Yao C, Gabillard D, Daures M, Augier A, Anglaret X, Kinda M, Shepherd S, Becquet R. Optimising the dosage of ready-to-use therapeutic food in children with uncomplicated severe acute malnutrition in the Democratic Republic of the Congo: a non-inferiority, randomised controlled trial. EClinicalMedicine. 2023 Feb 28;58:101878. doi: 10.1016/j.eclinm.2023.101878. eCollection 2023 Apr. PMID 36915287
- [Background] Bailey J, Opondo C, Lelijveld N, Marron B, Onyo P, Musyoki EN, Adongo SW, Manary M, Briend A, Kerac M. A simplified, combined protocol versus standard treatment for acute malnutrition in children 6-59 months (ComPAS trial): A cluster-randomized controlled non-inferiority trial in Kenya and South Sudan. PLoS Med. 2020 Jul 9;17(7):e1003192. doi: 10.1371/journal.pmed.1003192. eCollection 2020 Jul. PMID 32645109
- [Background] Isanaka S, Menzies NA, Sayyad J, Ayoola M, Grais RF, Doyon S. Cost analysis of the treatment of severe acute malnutrition in West Africa. Matern Child Nutr. 2017 Oct;13(4):e12398. doi: 10.1111/mcn.12398. Epub 2016 Dec 5. PMID 27921381
- [Background] Thompson DS, McKenzie K, Opondo C, Boyne MS, Lelijveld N, Wells JC, Cole TJ, Anujuo K, Abera M, Berhane M, Koulman A, Wootton SA, Kerac M, Badaloo A; CHANGE Study Collaborators Group. Faster rehabilitation weight gain during childhood is associated with risk of non-communicable disease in adult survivors of severe acute malnutrition. PLOS Glob Public Health. 2023 Dec 21;3(12):e0002698. doi: 10.1371/journal.pgph.0002698. eCollection 2023. PMID 38127945
- [Background] Olofin I, McDonald CM, Ezzati M, Flaxman S, Black RE, Fawzi WW, Caulfield LE, Danaei G; Nutrition Impact Model Study (anthropometry cohort pooling). Associations of suboptimal growth with all-cause and cause-specific mortality in children under five years: a pooled analysis of ten prospective studies. PLoS One. 2013 May 29;8(5):e64636. doi: 10.1371/journal.pone.0064636. Print 2013. PMID 23734210
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] McDonald CM, Olofin I, Flaxman S, Fawzi WW, Spiegelman D, Caulfield LE, Black RE, Ezzati M, Danaei G; Nutrition Impact Model Study. The effect of multiple anthropometric deficits on child mortality: meta-analysis of individual data in 10 prospective studies from developing countries. Am J Clin Nutr. 2013 Apr;97(4):896-901. doi: 10.3945/ajcn.112.047639. Epub 2013 Feb 20. PMID 23426036